CLINICAL TRIAL: NCT05658224
Title: Education Time Influence on Exercise-Induced Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Kory Zimney, PT, DPT, PhD, Associate Professor, University of South Dakota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: USouthDakota
Record Dates: First submitted 2022-11-30; First posted 2022-12-20 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Exercise
Keywords: Exercise induced hypoalgesia; Education
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized into 1 of 2 groups. Outcome assessor will not be informed of participant grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short education (Active Comparator): Individuals receiving a short (1-minute) educational session on exercise-induced hypoalgesia
  Interventions: Behavioral: Education on effects of Exercise-induced hypoalgesia from exercise
- Long education (Active Comparator): Individuals receiving long (10-15 minutes) educational session on exercise-induced hypoalgesia
  Interventions: Behavioral: Education on effects of Exercise-induced hypoalgesia from exercise

INTERVENTIONS:
Behavioral: Education on effects of Exercise-induced hypoalgesia from exercise — Educational session with participants

SUMMARY:
We will investigate the effects of the length of education on exercise-induced hypoalgesia (EIH). Two previous studies have shown that positive education about the effects of exercise and the phenomena of EIH produce enhancements to EIH response (having decreased reports of pain with exercise). These previous studies used different amounts of education time, this study will compare directly if the length of education time varies the effects on EIH.

DETAILED DESCRIPTION:
The use of fliers will be posted on USD campus explaining study and the need for volunteers. Potential volunteers will contact study personal listed on the flier to set up potential time for study enrollment. When the prospective participant arrives, they will be provided a hard copy of informed consent and study personnel will be available to answer questions. If the participant consents and signs, they will then be screened to ensure inclusion/exclusion by answering screening questions.

Once they have consented and met study inclusion/exclusion the participants will then be randomized into 1 of 2 groups by picking a number out of an envelope. Group 1 will receive a more extensive education session (10-15 min) on the benefits of exercise and EIH. Group 2 will receive a brief education session (1 minute) on the benefits of exercise and EIH. Next participants will complete basic demographic information: age, gender, history of injuries, athletic participation history, and Knowledge and Beliefs about Exercise and Pain Questionnaire (questions 1 -4).

Then they will be introduced and tested for pain pressure threshold (PPT). This standard measurement assesses the threshold when a pressure applied to the body passes from pressure to pain. A PPT algometer with a 1 cm tip is used to apply pressure to a body part slowly. When the participant first feels the sensation of pain, the pressure being applied is stopped and the amount of force is recorded as the individual's PPT. The participant will initially be introduced to the testing at the web space of the thumb and index finger on their dominant hand, this is done 3 times with minimum 15 seconds between each measurement and the average of the 3 measurements is used.

Participants then will receive the education about EIH depending on their group allocation last 1 minute or 10-15 minutes. After the education, the participants will be asked question #5 on the Knowledge and Beliefs about exercise and pain questionnaire. Both groups will be shown a picture of the exercise (wall squat) that they will perform and provided instruction on the exercise before they begin. The wall squat exercise will consist of standing upright with their back against the wall with feet 45 cm from the wall, feet parallel and shoulder width apart, and hands at their side. They will slide down the wall bending at the hips and knees, keeping their back against the wall and feet in place until their knee joint angle reaches 100 degrees of flexion measured by the study personnel. All participants are asked to maintain the position for 3 minutes or until fatigued and need to stop.

Prior to beginning the wall squat exercise, participants are asked to rate the intensity of pain in their legs using the Numeric Rating Scale (NRS=0-10, 0=no pain, 10=worst imaginable pain). Pain Pressure Threshold will be measured on the dominant quadriceps muscle and the non-dominate upper trapezius muscle. During the exercise, the NRS and category-ration scale of Rating of Perceived Exertion (CR 10, 0=nothing at all, 10=extremely strong) will be measured while performing the exercise at 1 minute, 2 minutes, and 3 minutes. Immediately post-exercise, Pain Pressure Threshold will be measured again on the dominant quadriceps muscle and the non-dominate upper trapezius muscle. The participants will also be asked to assess exercise expectations on EIH immediately post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand English,
* Refrained from alcohol, pain medication, and vigorous exercise for the past 24 hours,
* No history of chronic pain (pain > 3 months), or current pain/injury that would prevent the ability to do exercise.

Exclusion Criteria:

* unable to meet screening questions for PAR-Q+ for safe exercise

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kory Zimney, DPT, PT, Principal Investigator — University of South Dakota
Locations (1):
- University of South Dakota, Vermillion, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of study for 3 years after closing study.
Access Criteria: email PI at kory.zimney@usd.edu for data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Education | Long Education
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Education | Long Education | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (.837) | 24.2 (.837) | 24 (.775)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pain Pressure Threshold
Description: Measurement in kg/cm2, higher score is better outcome
Time Frame: 3 minutes post exercise on Day following educational session and exercise
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Short Education | Long Education
Number analyzed (Participants) | 5 | 5
kg/cm^2 | 0.72 (0.58) | 1.13 (2.39)

2. Secondary Outcome: Knowledge and Beliefs About Exercise and Pain Questionnaire
Description: paper questionnaire on Likert scale 1 strongly disagree, 5 strongly agree. higher number indicates more knowledge.
Time Frame: 3 minutes post exercise on Day following educational session and exercise
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Short Education | Long Education
Number analyzed (Participants) | 5 | 5
units on a scale | 3.4 (1.517) | 3.2 (.837)

ADVERSE EVENTS:
Time Frame: Participants were assessed during the intervention of the exercise protocol (3 imuntes) and for a follow-up of 10 minutes post exercise, they were to report any changes that may be due to adverse event for 3 days post exercise.
Arm/Group | Short Education | Long Education
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT05658224/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT05658224/ICF_001.pdf